CLINICAL TRIAL: NCT06143072
Title: Referral Pathways and Care Provision for Patients Who Develop OASI Associated Incontinence in the First Five Years Following a Vaginal Delivery
Brief Title: CArE for OAsI Study: Care Pathways and Anorectal Evaluation for OASI Associated Incontinence
Acronym: CArE for OAsI
Status: Recruiting | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 333989
Record Dates: First submitted 2023-11-06; First posted 2023-11-22 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Obstetric Anal Sphincter Injury; Severe Perineal Trauma; Grade 3 Perineal Tear; Grade 4 Perineal Tear; Anal Incontinence; Faecal Incontinence; Urgency; Deferral Time; Pathways; Follow-up; Review; Endo-anal Ultrasound; Urogynaecology; Biofeedback
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part 1 of study: Women who have sustained an obstetric-related anal sphincter injury (grade 3 and 4 perineal tears) AND who are symptomatic of anal/faecal incontinence within the first five years following a vaginal delivery are eligible to participate, provided they have capacity to consent.
- Part 2 of study: Obstetricians (consultants) and urogynaecologists who are involved in and/or oversee the care of OASI patients' post-partum in the UK.

SUMMARY:
The aim of this study is to ascertain which pathways currently exist in relation to the follow up of patients with obstetric anal sphincter injury related incontinence. This is particularly important as afflicted individuals may not readily volunteer information about their symptoms and struggles and need to be safeguarded by the presence of robust care pathways that ensure adequate follow up and care provision.

As obstetric anal sphincter injuries have been associated with increased litigation rates over the years, positive interventions towards patient care will help ameliorate the financial burden that litigation carries on the National Health Service. It is noteworthy of mention that perineal injury, in itself, may not be suggestive of negligent care and is a recognized complication of vaginal delivery. However, a failure to adequately manage the injury may carry medicolegal implications.

DETAILED DESCRIPTION:
Historically, pregnancy and childbirth has been erroneously considered to be an innocuous physiological event. However, vaginal delivery may be associated with perineal injury, a common occurrence affecting up to 80% of women. Perineal injury is classified into four categories, as per the Sultan classification:

Grade 1: involvement of perineal skin +/- vaginal mucosa Grade 2: involvement of perineal muscles Grade 3a: <50% External Anal Sphincter (EAS) Grade 3b: >50% EAS Grade 3c: EAS + Internal Anal Sphincter (IAS) Grade 4: Grade 3c + anorectal mucosa The latter two categories are associated with considerable morbidity and are known as obstetric anal sphincter injuries (OASIS). OASIS encompass grade 3 and 4 perineal tears and effect the integrity of the anorectal sphincter complex, with or without involvement of the anorectal mucosa.

Such injuries may be associated with a myriad of devastating and stigmatizing sequelae, including faecal and urinary incontinence, dyspareunia, rectovaginal fistulae, perineal pain and pelvic organ prolapse, which in turn may have a negative impact on a woman's quality of life and day-to-day living. Indeed, sustaining an Obstetric Anal Sphincter Injury (OASI) has been associated with both physical and psychological sequelae.

Symptoms of urgency and urge faecal incontinence, are suggestive of damage to the external anal sphincter, while symptoms of passive leakage are indicative of damage to the internal anal sphincter. Not all women with OASIS are symptomatic. Symptomatic OASIS occurs in about 30-50% of women. It is important to note that the real incidence may be higher as it may very well be underreported.

The incidence of OASIS in the UK is 2.9%. Although OASIS is uncommon, the rate of OASIS in singleton, cephalic and first vaginal deliveries, has reportedly tripled from 1.8% to 5.9% from 2000 to 2012. This may, however, be secondary to better detection of these injuries following improvements in education, training and the utilization of a standardized classification system for perineal tears. To address the rising OASI rates, the OASI care bundle was introduced which primarily focused on interventions in the antenatal period to reduce the incidence of OASIS. Prevention of OASIS, however, will not always be possible, even with the best efforts of care. Therefore, focus should also be placed on the optimal management of these patients' post-partum.

The RCOG (royal college of obstetricians and gynaecologists) guidance states that clinicians should diagnose an OASI at the time of delivery by meticulous inspection of the perineum, which should include a digital rectal examination. Referral to a colorectal specialist should be considered in those who are symptomatic of incontinence. However, in the absence of a standardised national pathway, the provision of healthcare appears to rely heavily on the availability of resources, a clinician's discretion and ultimately a 'postcode lottery'. Indeed, while some trusts may have the necessary provisions in place to support mothers with OASIS, in other areas, women may be left to fend for themselves.

Moreover, the stigma and shame associated with sustaining such an injury may perpetuate the difficulty in seeking medical attention, even in the most motivated patients, thereby producing a population of silent sufferers, who are stuck in a pervasive pattern of shame, embarrassment and inevitably, melancholy.

There may also be the erroneous belief among healthcare professionals, that these symptoms would settle on their own and this may be communicated to the afflicted individual who may be reassured by this information. Although 60-80% of women are asymptomatic at one year, some remain symptomatic, with devastating consequences on their quality of life. Further, patients with an asymptomatic injury ought to be counselled regarding the risk of incontinence in later life, secondary to advancing age and hormonal influence on pelvic floor function as well as the added impact of future deliveries. When discussing mode of delivery for future pregnancies, it should be highlighted that although an elective caesarean section may protect against an anal sphincter injury, it may not prevent pudendal neuropathy which may also contribute to symptoms of incontinence.

ELIGIBILITY:
Part 1 of Study

Inclusion Criteria:

* • Fertile women ≥ 18 years and ≤50 who have developed OASI related incontinence following a vaginal delivery in the preceding five years (N.B. the average age of menopause in the UK is 51)

  * Tertiary referrals to the specialist perineal clinic as well as patients who have 'slipped' through the existing pathway of referral
  * Capacity to consent (able to comprehend and retain information, weight out the risks and benefits and communicate a decision back to the researcher)
  * English-speaking and able to comprehend and read English
  * Primiparous/multi-parous

Exclusion Criteria:

* • Women who are unable to consent or who have severe mental illness, as decided by the screening clinician

  * Patients who do not speak, read or understand English
  * Patients with an alternative documented cause for their FI that is non obstetric trauma related.
  * Post-menopausal women who may develop late onset symptoms of incontinence relating to a previous OASI (clinically silent injuries that manifest in later life secondary to hormonal influences or advancing age for example).
  * Women with an OASI who have been referred directly from the maternity unit at the same trust as the specialist perineal clinic, where an existing trust policy exists for direct referral of these patients from the maternity unit to the perineal clinic.

Part 2 of study:

Inclusion criteria:

• urogynaecologists/obstetricians who oversee the care of or look after patients with OASI and who are practising in UK NHS hospitals at the time of completion of the survey. They must be on the GMC specialist register to be eligible to participate

Exclusion criteria:

• trainees, obstetricians/gynaecologists not routinely involved in the care of OASI patients.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: There are two parts to study:
  Part 1: semi-structured interview, retrospective study, mix of qualitative and quantitative methods - involving patients. Women who have sustained an obstetric-related anal sphincter injury (grade 3 and 4 perineal tears) AND who are symptomatic of anal/faecal incontinence within the first five years following a vaginal delivery are eligible to participate, provided they have capacity to consent.
  Part 2: Cross-sectional, observational study with a mix of qualitative and quantitative analysis, using a survey, to be completed by urogynaecologists/obstetricians Obstetricians (consultants) and urogynaecologists who are involved in and/or oversee the care of OASI patients' post-partum in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The patient's perception of the quality of care received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering whether the patient was assessed clinically for incontinence during the post-partum check at 6-12 weeks conducted by the obstetrics/urogynaecology team (part 1 of study)
The patient's perception of the quality of care received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering the ease with which they were able to discuss the symptoms of incontinence with a clinician (part 1 of study)
The patient's perception of the quality of care received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering how symptoms were managed before consulting a clinician and after (part 1 of study)
The patient's perception of the quality of care received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering who they saw during their follow up appointments and when (including referrals), and what was discussed and what action was taken for the management of their incontinence (including counselling regarding future pregnancies) (part 1 of study)
The Obstetrics and Urogynaecologists perception of the quality of care the patient has received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering whether the patient was assessed clinically for incontinence during the post-partum check at 6-12 weeks as conducted by the team (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care the patient has received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering how these patients are assessed (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care the patient has received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering the length of time taken to follow up a patient (whether symptomatic or asymptomatic) (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care the patient has received following OASI-associated incontinence, as a measure of follow up care | 12 months
  considering if there is a policy/pathway in place for the management of OASI-associated incontinence (part 2 of study)

SECONDARY OUTCOMES:
Degree of OASI in relation to symptoms and Quality of Life, evaluated using a patient's own verbatim account of their lived experience and assessed via open ended questions in a semi-structured interview. | 12 months
  The influence of severity of OASI on incontinence, and the latter's effect on the patient's quality of life (including effect on job, family and relationships) (part 1 of study)
The Obstetrics and Urogynaecologists perception of the quality of care received following OASI-associated incontinence, as a measure of being seen/reviewed by other members of the MDT | 12 months
  considering: whether or not these patients are discussed in the MDT (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care received following OASI-associated incontinence, as a measure of being seen/reviewed by other members of the MDT | 12 months
  considering whether or not these patients are reviewed by a physiotherapist and if so, at what stage post-partum? (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care received following OASI-associated incontinence, as a measure of being seen/reviewed by other members of the MDT | 12 months
  considering: If they are referred for anorectal studies (part 2 of study)
The Obstetrics and Urogynaecologists perception of the quality of care received following OASI-associated incontinence, as a measure of being seen/reviewed by other members of the MDT | 12 months
  considering whether or not these patients are referred for biofeedback and if not, why. (part 2 of study)

CONTACTS AND LOCATIONS:
Locations (1):
- London Northwest Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No